CLINICAL TRIAL: NCT01410084
Title: Improving Vitamin D Status in Home-bound Elders: a Pilot Study
Brief Title: Improving Vitamin D Status in Home-bound Elders
Acronym: MOW VitD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014152
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-07

CONDITIONS: Vitamin D Deficiency; Accidental Falls
Keywords: vitamin D; falls; deficiency; insufficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin E

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 (Experimental): 100,000 IU vitamin D3 once monthly
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin E (Placebo Comparator): 400 IU vitamin E once monthly
  Interventions: Dietary Supplement: Vitamin E

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 100,000 IU vitamin D3 once monthly for 5 months
  Arms: Vitamin D3
Dietary Supplement: Vitamin E — 400 IU vitamin E once monthly for 5 months
  Arms: Vitamin E

SUMMARY:
In the past two decades, the role of vitamin D has extended beyond bone health to encompass a wide range of biological activities important to physical function in older adults. A growing body of evidence now shows that circulating 25-hydroxyvitamin D (25(OH)D) levels < 75 nmol/L (< 30 ng/mL)) are associated with physical impairments such as reduced walking speed and impaired balance as well as falls. Older adults are at risk for low levels of 25-hydroxyvitamin D because of reduced exposure to ultraviolet B radiation, reduced efficiency of previtamin D synthesis in the skin, and low dietary intake. Although data from the National Health and Nutrition Examination Survey (NHANES) 2000-2004 indicate that frank vitamin D deficiency (serum 25(OH)D < 25 nmol/L [10 ng/mL]) is rare in the U.S. (5% or less), vitamin D insufficiency (serum 25(OH)D < 75 nmol/L [30 ng/mL]) is prevalent (~75%) among older adults. Older home-bound adults are a vulnerable subgroup of older adults for poor dietary intake and nutritional health, nutrition-related health conditions, and functional decline and disability. The primary goal of this pilot study is to assess the feasibility of a partnership with Senior Services of Forsyth County to address vitamin D insufficiency in home-bound older adults receiving home-delivered meals. A secondary goal is to obtain preliminary data on the effectiveness of vitamin D supplementation on improving vitamin D levels and reducing falls.

DETAILED DESCRIPTION:
In the past two decades, the role of vitamin D has extended beyond bone health to encompass a wide range of biological activities important to physical function in older adults. A growing body of evidence now shows that circulating 25-hydroxyvitamin D (25(OH)D) levels < 75 nmol/L (< 30 ng/mL)) are associated with physical impairments such as reduced walking speed and impaired balance as well as falls. Older adults are at risk for low levels of 25-hydroxyvitamin D because of reduced exposure to ultraviolet B radiation, reduced efficiency of previtamin D synthesis in the skin, and low dietary intake. Although data from the National Health and Nutrition Examination Survey (NHANES) 2000-2004 indicate that frank vitamin D deficiency (serum 25(OH)D < 25 nmol/L [10 ng/mL]) is rare in the U.S. (5% or less), vitamin D insufficiency (serum 25(OH)D < 75 nmol/L [30 ng/mL]) is prevalent (~75%) among older adults. Older home-bound adults are a vulnerable subgroup of older adults for poor dietary intake and nutritional health, nutrition-related health conditions, and functional decline and disability. The primary goal of this pilot study is to assess the feasibility of a partnership with Senior Services of Forsyth County to address vitamin D insufficiency in home-bound older adults receiving home-delivered meals. The investigators will accomplish this goal by conducting a 5-month randomized, controlled trial in 200 older Meals-on-Wheels (MOW) recipients randomized to receive monthly either (1) 100,000 IU vitamin D3 or (2) an active placebo (vitamin E) to achieve the following specific aims:

Aim 1: Determine the prevalence of falls and risk of vitamin D insufficiency in 200 MOW recipients.

Aim 2: Assess the feasibility of the vitamin D intervention delivered through the MOW program.

Aim 3: Obtain preliminary data on the effectiveness of the intervention on improving vitamin D status and reducing falls.

Data from this pilot study will: 1) provide estimates of the prevalence of falls and vitamin D insufficiency in home-bound older adults participating in the Forsyth County MOW program; 2) provide estimates of participant compliance and drop-out to a vitamin supplementation trial delivered as part of the MOW program; 3) provide evidence for the efficacy of the vitamin D dose proposed in remediating vitamin D insufficiency; and 4) provide preliminary data on the potential benefit of vitamin D supplementation on falls in a home-bound older population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old
* Forsyth County Senior Services Meals-on-Wheels recipient
* Willing to provide informed consent
* Willing to be randomized to vitamin D or active placebo control

Exclusion Criteria:

* Hyperparathyroidism
* Kidney stones (within the past 2 years)
* History of hypercalcemia
* On dialysis
* Inability or contraindications to consume vitamin D supplements
* Taking prescription vitamin D2 or vitamin D3-containing supplements totaling > 1000 IU/d
* Planning to move within the next 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise K Houston, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D3 | Vitamin E
Started | 38 | 30
Completed | 37 | 27
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 | Vitamin E | Total
Number analyzed (Participants) | 38 | 30 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 38 | 30 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (9.0) | 78.2 (8.4) | 77.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 19 | 49
  Male | 8 | 11 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 24 | 51
  White | 11 | 6 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in 25-hydroxyvitamin D Levels Over 5 Months
Description: Determine the effectiveness of the intervention on improving 25-hydroxyvitamin D levels (change in 25(OH)D from baseline to 5-month follow-up). Measured as 5-month follow-up 25(OH)D level minus baseline 25(OH)D level.
Time Frame: 5 months
Population: Participants who did not have a 5 month follow-up visit (n=4) and those who did not have baseline and/or follow-up blood samples (n=7) were excluded from the analysis leaving an analysis sample of 57 participants
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Vitamin D3 | Vitamin E
Number analyzed (Participants) | 33 | 24
ng/mL | 21.7 (3.1) | 0 (4.0)

2. Secondary Outcome: Number of Falls
Description: Determine the effectiveness of the intervention on reducing the number of falls using monthly fall calendars (compare the average number of falls in vitamin D3 group vs. active placebo group over 5 months)
Time Frame: 5 months
Measure: Mean (Full Range); unit: falls/participant
Arm/Group | Vitamin D3 | Vitamin E
Number analyzed (Participants) | 33 | 26
falls/participant | 0.5 [0 to 4] | 1.1 [0 to 8]

3. Secondary Outcome: Number of Participants Who Were Compliant to Intervention
Description: Number of participants who consumed at least 4 out of a possible 5 supplement doses (=>80% compliance) over 5 months.
Time Frame: 5 months
Population: Compliance assessed in participants who remained in the study over the 5 month intervention for an analysis sample of 64 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 | Vitamin E
Number analyzed (Participants) | 37 | 27
Participants | 37 | 24

ADVERSE EVENTS:
Arm/Group | Vitamin D3 | Vitamin E
All-Cause Mortality (participants affected / at risk) | 0/38 | 3/30
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/30
Other Adverse Events (participants affected / at risk) | 0/38 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No